CLINICAL TRIAL: NCT05627024
Title: Effects of Different Inhalation Oxygen Concentrations on Oxygenation Index and Immediately Postoperative Atelectasis in Neurosurgery Patients. DIOCA-Trial
Brief Title: Effects of Different Inhalation Oxygen Concentrations on Postoperative Atelectasis
Acronym: DIOCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-381
Record Dates: First submitted 2022-11-14; First posted 2022-11-25 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In addition to the anesthesiologist on the day of surgery, the patients and all participants, statistical analysts, ward staff, surgeons, and treatment-outcome assessors are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 30% Oxygen (Experimental): Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 mins. After successful anesthesia induction, Fio2 will be adjusted to 30%, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cmh2O, RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation, however when intraoperative oxygen saturation is less than 92% the manual lung recruitment maneuver will be done too. Arterial blood will be collected twice for blood gas analysis, the first once is in the non-oxygen inhalation state before anesthesia induction and the second is 30min before the end of surgery. Patients in both groups will be extubated in the operating room and then sent to the PACU.
  Interventions: Drug: 30% Oxygen
- Placebo Comparator: 60% Oxygen (Placebo Comparator): Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 mins. After successful anesthesia induction, Fio2 will be adjusted to 60%, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cmh2O, RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Arterial blood will be collected twice for blood gas analysis, the first once is in the non-oxygen inhalation state before anesthesia induction and the second is 30min before the end of surgery. Patients in both groups will be extubated in the operating room and then sent to the PACU.
  Interventions: Drug: 60% Oxygen

INTERVENTIONS:
Drug: 30% Oxygen — Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 mins. After successful anesthesia induction, Fio2 will be adjusted to 30%, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cmh2O, RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation, however when intraoperative oxygen saturation is less than 92% the manual lung recruitment maneuver will be done too. Arterial blood will be collected twice for blood gas analysis, the first once is in the non-oxygen inhalation state before anesthesia induction and the second is 30min before the end of surgery. Patients in both groups will be extubated in the operating room and then sent to the PACU.
  Arms: Experimental: 30% Oxygen
Drug: 60% Oxygen — Before anesthesia induction, the participants inhaled pure oxygen through the mask for 5 mins. After successful anesthesia induction, Fio2 will be adjusted to 60%, and the total gas flow rate will be set at 2L/min. All patients will be performed via the lung protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cmh2O, RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Arterial blood will be collected twice for blood gas analysis, the first once is in the non-oxygen inhalation state before anesthesia induction and the second is 30min before the end of surgery. Patients in both groups will be extubated in the operating room and then sent to the PACU.
  Arms: Placebo Comparator: 60% Oxygen

SUMMARY:
This study was a single-center, prospective, randomized controlled, two-arm study. This study will be conducted in the First Hospital of China Medical University. the investigators aimed to investigate the effects of different inspired oxygen concentrations in lung protective ventilation strategies on immediate postoperative atelectasis and intraoperative changes of oxygenation index in patients undergoing neurosurgical surgery in the supine position.

DETAILED DESCRIPTION:
This study was a single-center, prospective, randomized controlled, two-arm study. This study will be conducted in the First Hospital of China Medical University. the investigators aimed to investigate the effects of different inspired oxygen concentrations in lung protective ventilation strategies on immediate postoperative atelectasis and intraoperative changes of oxygenation index in patients undergoing neurosurgical surgery in the supine position. A total of 96 neurosurgical patients under supine position were selected with an estimated operation time of more than 2 hours. Patients were randomly assigned to low-oxygen concentration (30%FiO2) L group, or high-oxygen concentration (60%FiO2) H group, and both groups received lung protective ventilation strategies. The main outcome was the comparison of postoperative atelectasis volume between the two groups. Secondary outcomes were the comparison of intraoperative oxygenation index and postoperative changes in diaphragm height between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologist (ASA) physical status I-II;
* Older than 18 years; Patients with operation time more than 2 hours and plan to extubate in the operating room;
* Preoperative blood gas partial pressure of oxygen was more than 80mmHg;
* Patients scheduled for elective neurosurgery were operated in the supine position.

Exclusion Criteria:

* A history of acute lung injury with acute respiratory distress syndrome within three months;
* Heart failure (New York Heart Association class) greater than IV, severe liver and kidney dysfunction (Child B or C liver failure, glomerular filtration rate <30ml/min);
* BMI > 30 kg/m2.
* The operation time is more than 10 hours;
* The amount of bleeding was more than 500ml; The total fluid volume exceeded 3000ml.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
the occurrence of atelectasis | On the operating room within 40 minutes after awakening
  The primary outcome is the occurrence of atelectasis scanned by computerized tomography in the operating room within 40 minutes after awakening.

SECONDARY OUTCOMES:
oxygenation index | On the operating room within 40 minutes after awakening
  The secondary outcome is the comparison of the oxygenation index between the two groups, which is calculated and compared from the results of intraoperative blood gas analysis.
bilateral diaphragmatic muscles | On the operating room within 40 minutes after awakening
  By comparing the preoperative and postoperative lung CT, the distance between the two lungs to the bilateral diaphragmatic muscles will be calculated and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided